CLINICAL TRIAL: NCT04085328
Title: Clinical Safety and Effectiveness Assessment of an Investigational Frequent Replacement Silicone Hydrogel Lens
Brief Title: Assessment of an Investigational Frequent Replacement Silicone Hydrogel Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLL949-C010
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-05

CONDITIONS: Refractive Ametropia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- LID015385 (Experimental): LID015385 soft contact lenses worn in both eyes for up to 6 nights/7 days continuously (awake and asleep). Must sleep 1 night per week without lenses. Lenses will be replaced as specified in the study protocol.
  Interventions: Device: LID015385 soft contact lenses
- Biofinity (Active Comparator): Comfilcon A soft contact lenses worn in both eyes for up to 6 nights/7 days continuously (awake and asleep). Must sleep 1 night per week without lenses. Lenses will be replaced as specified in the study protocol.
  Interventions: Device: Comfilcon A soft contact lenses

INTERVENTIONS:
Device: LID015385 soft contact lenses — Investigational silicone hydrogel contact lenses for up to 6 nights/7 days of continuous wear
  Arms: LID015385
Device: Comfilcon A soft contact lenses — Silicone hydrogel contact lenses for up to 6 nights/7 days of continuous wear
  Other Names: BIOFINITY®
  Arms: Biofinity

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and performance of an investigational soft contact lens compared to a commercially available soft contact lens when worn in an extended wear modality.

DETAILED DESCRIPTION:
Subjects will be expected to attend 9 office visits. The total expected duration of participation for each subject is approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign an Informed Consent Form.
* Willing to attend all scheduled study visits as required per protocol.
* Willing and able to wear assigned study lenses as required per protocol.
* Successful wear of spherical daily wear or extended wear frequent replacement soft contact lenses in both eyes during the past 3 months for a minimum of 5 days per week.
* Manifest cylinder ≤ 0.75 diopter (D) in each eye.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Any eye infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the Investigator.
* Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the Investigator.
* History of eye surgery, including refractive surgery.
* Currently pregnant or breast-feeding.
* Monovision contact lens wearers.
* Daily disposable contact lens wearers.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alcon Study Director, Study Director — Alcon Research
Locations (42):
- United States (42):
  - Family EyeCare Center, Campbell, California
  - Winston Eye Care, Fullerton, California
  - Kurata Eye Care Center, Los Angeles, California
  - East West Eye Institute, Los Angeles, California
  - Dr.Elsa Pao, O.D, Oakland, California
  - Gordon Schanzlin New Vision Institute, San Diego, California
  - Complete Family Vision Care, San Diego, California
  - Westview Optometry, San Diego, California
  - OMEGA Vision Center PA, DBA Sabal Eye Care, Longwood, Florida
  - Kindred Optics at Maitland Vision Center, Maitland, Florida
  - Mid Florida Eye Center, PA, Mt. Dora, Florida
  - Eola Eyes, Orlando, Florida
  - Vision Health Institute, Orlando, Florida
  - Visual Performance Center Research & Development, Pensacola, Florida
  - Golden Vision, Sarasota, Florida
  - Advanced Eyecare Specialists, West Palm Beach, Florida
  - VisionPoint Eye Center, Bloomington, Illinois
  - Franklin Park Eye Center, PC, Franklin Park, Illinois
  - Kannarr Eye Care, LLC, Pittsburg, Kansas
  - Optimum Vision Care, Brighton, Massachusetts
  - Fraser Eye Care Center, Fraser, Michigan
  - Dr. Schwartz Optometrist and Associates, Sterling Heights, Michigan
  - Complete Eye Care of Medina, Medina, Minnesota
  - Fischer Laser Eye Center, LLC, Willmar, Minnesota
  - Tekwnai Vision Center, Inc, St Louis, Missouri
  - Alterman, Modi & Wolter, Poughkeepsie, New York
  - Rochester Ophthalmological Group, PC, Rochester, New York
  - Asheville Eye Associates, PLLC, Asheville, North Carolina
  - ProCare Vision Centers, Inc., Granville, Ohio
  - Midwest Vision Care, Piqua, Ohio
  - EyeCare Professionals, Inc. DBA Insight Research Clinic, LLC, Powell, Ohio
  - Wyomissing Optometric Center, Wyomissing, Pennsylvania
  - West Bay Eye Associates, Warwick, Rhode Island
  - North Spartanburg Eye Center, Boiling Springs, South Carolina
  - Primary Eyecare Group, PC, Brentwood, Tennessee
  - Optometry Group, PLLC, Memphis, Tennessee
  - Total Eye Care, PA, Memphis, Tennessee
  - Advancing Vision Research, LLC, Smyrna, Tennessee
  - Beaumont Family Eye Care, Beaumont, Texas
  - Vision One Eyecare, Katy, Texas
  - Dawn M Rakich, OD, San Antonio, Texas
  - Clarke EyeCare Center, Wichita Falls, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population consisted of a Primary cohort, including subjects of any race/ethnic background at 35 Primary cohort sites, and a Supplemental cohort, including subjects of Chinese race only at 7 Supplemental cohort sites.
Pre-assignment Details: Of the 675 enrolled, 30 participants were exited from the study as screen failures prior to randomization. This reporting group includes all enrolled and dispensed participants (645).
Units Other Than Participants: eyes
Groups:
- Biofinity: Comfilcon A soft contact lenses worn in both eyes for up to 6 nights/7 days continuously (awake and asleep). Must have slept 1 night per week without lenses. Lenses were replaced as specified in the study protocol.
- LID015385: LID015385 soft contact lenses worn in both eyes for up to 6 nights/7 days continuously (awake and asleep). Must have slept 1 night per week without lenses. Lenses were replaced as specified in the study protocol.
Period: Overall Study
Arm/Group | Biofinity | LID015385
Started (Includes Primary Cohort and Supplemental Cohort) | 323; 646 eyes | 322; 644 eyes
Primary Cohort Started | 291; 582 eyes | 290; 580 eyes
Primary Cohort Completed | 256; 512 eyes | 257; 514 eyes
Primary Cohort Discontinued | 35; 70 eyes | 33; 66 eyes
Completed (Includes Primary Cohort and Supplemental Cohort) | 285; 570 eyes | 286; 572 eyes
Not Completed | 38; 76 eyes | 36; 72 eyes
Not completed — Witihdrew Consent | 16 | 16
Not completed — Adverse Event | 8 | 7
Not completed — Lost to Follow-up | 7 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Reasons Related to COVID-19 | 5 | 8
Not completed — Did not meet inclusion criteria | 1 | 1
Not completed — Early termination | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes enrolled subjects who were also dispensed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Biofinity | LID015385 | Total
Number analyzed (Participants) | 323 | 322 | 645
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (8.3) | 34.2 (9.5) | 33.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 197 | 399
  Male | 121 | 125 | 246
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 32 | 60
  Not Hispanic or Latino | 295 | 289 | 584
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 35 | 35 | 70
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 15 | 37
  White | 254 | 262 | 516
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 323 | 322 | 645

OUTCOME MEASURES:

1. Primary Outcome: Distance Visual Acuity (VA) With Study Lenses - Completed Eyes
Description: Visual acuity (VA) was assessed for each eye individually with study lenses in place at a distance of 6 meters using a letter chart. VA was collected in Snellen and converted to logarithm minimum angle of resolution (logMAR). A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with lower logMAR values indicating better visual acuity. No formal hypothesis was formulated for the primary effectiveness endpoint of distance VA; hence, no inferential testing was performed.
Time Frame: Day 1 Dispense; Hour 24 Follow-Up; Week 1 Follow-up; Month 1 Follow-up; Month 2 Follow-up; Month 3 Follow-up; Month 6 Follow-up; Month 9 Follow-up, Month 12 Follow-up
Population: This analysis population includes all enrolled dispensed subjects/eyes completing the study, with data at scheduled study visit. This outcome measure was pre-specified for the Primary Cohort.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Biofinity | LID015385
Number analyzed (Participants) | 256 | 257
Number analyzed (eyes) | 512 | 514
logMAR
  Day 1 Dispense | -0.05 (0.06) | -0.05 (0.06)
  Hour 24 Follow-up | -0.05 (0.06) | -0.05 (0.07)
  Week 1 Follow-up: number analyzed (Participants) | 254 | 252
  Week 1 Follow-up: number analyzed (eyes) | 508 | 504
  Week 1 Follow-up | -0.05 (0.06) | -0.05 (0.07)
  Month 1 Follow-up: number analyzed (Participants) | 240 | 236
  Month 1 Follow-up: number analyzed (eyes) | 480 | 472
  Month 1 Follow-up | -0.05 (0.07) | -0.05 (0.06)
  Month 2 Follow-up: number analyzed (Participants) | 234 | 237
  Month 2 Follow-up: number analyzed (eyes) | 468 | 474
  Month 2 Follow-up | -0.06 (0.06) | -0.05 (0.06)
  Month 3 Follow-up: number analyzed (Participants) | 244 | 242
  Month 3 Follow-up: number analyzed (eyes) | 488 | 484
  Month 3 Follow-up | -0.06 (0.07) | -0.05 (0.06)
  Month 6 Follow-up: number analyzed (Participants) | 253 | 254
  Month 6 Follow-up: number analyzed (eyes) | 506 | 508
  Month 6 Follow-up | -0.06 (0.06) | -0.06 (0.06)
  Month 9 Follow-up: number analyzed (Participants) | 253 | 257
  Month 9 Follow-up: number analyzed (eyes) | 506 | 514
  Month 9 Follow-up | -0.06 (0.06) | -0.05 (0.06)
  Month 12 Follow-up/Exit | -0.06 (0.06) | -0.05 (0.07)

2. Primary Outcome: Distance Visual Acuity (VA) With Study Lenses - Discontinued Eyes
Description: as for outcome 1
Time Frame: Day 1 Dispense; Hour 24 Follow-Up; Week 1 Follow-up; Month 1 Follow-up; Month 2 Follow-up; Month 3 Follow-up; Month 6 Follow-up; Month 9 Follow-up
Population: This analysis population includes all enrolled and dispensed subjects/eyes not completing the study, with data at scheduled study visit. This outcome measure was pre-specified for the Primary Cohort.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Arm/Group | Biofinity | LID015385
Number analyzed (Participants) | 35 | 33
Number analyzed (eyes) | 70 | 66
logMAR
  Day 1 Dispense | -0.04 (0.06) | -0.06 (0.07)
  Hour 24 Follow-up: number analyzed (Participants) | 31 | 32
  Hour 24 Follow-up: number analyzed (eyes) | 62 | 64
  Hour 24 Follow-up | -0.03 (0.06) | -0.05 (0.07)
  Week 1 Follow-up: number analyzed (Participants) | 26 | 27
  Week 1 Follow-up: number analyzed (eyes) | 52 | 54
  Week 1 Follow-up | -0.05 (0.06) | -0.05 (0.08)
  Month 1 Follow-up: number analyzed (Participants) | 21 | 21
  Month 1 Follow-up: number analyzed (eyes) | 42 | 42
  Month 1 Follow-up | -0.04 (0.06) | -0.05 (0.06)
  Month 2 Follow-up: number analyzed (Participants) | 19 | 12
  Month 2 Follow-up: number analyzed (eyes) | 38 | 24
  Month 2 Follow-up | -0.06 (0.06) | -0.04 (0.11)
  Month 3 Follow-up: number analyzed (Participants) | 17 | 9
  Month 3 Follow-up: number analyzed (eyes) | 34 | 18
  Month 3 Follow-up | -0.05 (0.06) | -0.02 (0.07)
  Month 6 Follow-up: number analyzed (Participants) | 10 | 5
  Month 6 Follow-up: number analyzed (eyes) | 20 | 10
  Month 6 Follow-up | -0.07 (0.06) | -0.07 (0.06)
  Month 9 Follow-up: number analyzed (Participants) | 4 | 2
  Month 9 Follow-up: number analyzed (eyes) | 8 | 4
  Month 9 Follow-up | -0.08 (0.06) | -0.12 (0.00)

3. Primary Outcome: Proportion of Ocular Serious and Significant Non-serious Adverse Device Effects (ADEs)
Description: Calculated as the total number of eyes reporting at least one treatment-emergent, ocular, serious ADE or treatment-emergent, ocular, significant, non-serious ADE, divided by the total number of eyes enrolled and dispensed. An ADE was defined as any adverse event related to the use of the investigational medical device (LID015385) or control product (Biofinity).
Time Frame: Up to Month 12
Population: This analysis population includes all enrolled subjects who were also dispensed. This outcome measure was pre-specified for the Primary Cohort.
Measure: Number; unit: proportion of eyes
Units Other Than Participants: eyes
Arm/Group | Biofinity | LID015385
Number analyzed (Participants) | 291 | 290
Number analyzed (eyes) | 582 | 580
proportion of eyes | 0.0258 | 0.0103
Statistical Analysis 1: Comparison: Biofinity vs LID015385; Test type: Non-Inferiority — Predefined margin of 0.05 for noninferiority; Generalized linear model; Proportion of events was analyzed using a generalized linear model, with a logit link function, accounting for within-subject correlation; Difference in proportion = -0.0154, 95% CI 1-sided [upper limit -0.0015] — Difference in proportion = LID015385 minus Biofinity

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 12 months.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. This analysis population includes all enrolled and dispensed subjects.
Groups:
- Pretreatment: Events reported in this group occurred prior to dispense of the study contact lenses
- Control Ocular; Control Nonocular: Events reported in this group occurred following dispense of the comfilcon A contact lenses
- Test Ocular; Test Nonocular: Events reported in this group occurred following dispense of the LID015385 contact lenses
Arm/Group | Pretreatment | Control Ocular | Control Nonocular | Test Ocular | Test Nonocular
All-Cause Mortality (participants affected / at risk) | 0/645 | 0/646 | 0/323 | 0/644 | 0/322
Serious Adverse Events (participants affected / at risk) | 0/645 | 4/646 | 2/323 | 0/644 | 3/322
Other Adverse Events (participants affected / at risk) | 0/645 | 0/646 | 0/323 | 0/644 | 0/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=645) | Control Ocular (N=646) | Control Nonocular (N=323) | Test Ocular (N=644) | Test Nonocular (N=322)
Ulcerative keratitis (Eye disorders) | 0 | 4 | 0 | 0 | 0
Hypopyon (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
Intervertebral disc operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/28/NCT04085328/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT04085328/SAP_001.pdf